CLINICAL TRIAL: NCT05283772
Title: Developing and Examining the Effectiveness of an Eye Tracker for Simulation Training in Nursing: A Double-blind Randomized Controlled Study
Brief Title: Developing and Examining the Effectiveness of an Eye Tracker for Simulation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Mehmet Halil Öztürk, Lecturer, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E-76261397-050.99-37648
Record Dates: First submitted 2022-02-17; First posted 2022-03-17 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Nursing Education; Eye Tracker; Simulation Training
Keywords: Nursing; Education; Eye tracker; Simulation
MeSH Terms: interventions — Nursing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: Development of eye tracker for simulation training in nursing
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Development of eye tracker for simulation training in nursing — Purpose: To develop a cost-effective and effective eye tracker for simulation training in nursing in Turkey.
  The wearable eye tracker consists of a front camera that will detect the pupil and determine the gaze region of the eye, and glasses or an alternative headband to which these cameras will be connected. A portable mini-computer will be used to process the obtained images. While recording and monitoring the eye movement with the pupil detection camera, real-world images in the user's field of view will be recorded by the front camera and the focal points will be determined. By establishing a linear connection between these found points, temperature (heat) maps will be created at the points where the eye looks.
  Arms: Experimental

SUMMARY:
Today, rapid developments in technology and science; affected the economic, cultural, political and social fields. The use of technology in these areas has become a necessity rather than a privilege. Education is one of the areas where technology is used the most and most intensely affected. Different education and training technologies can be used at every stage of the education and training process. With the effective and correct use of technology, it is possible to provide efficient and effective service in the fields of education and health care. This situation is gaining more and more importance for our country in the fields of nursing practice and education. Nursing organizations accept technology as the basic building block of nursing education and practice. Simulation is defined as "a technique of developing real patient experiences and the most important aspects of the real world from experience using practice guides in a completely interactive way". According to the World Health Organization, the use of simulation methods for teaching and learning is one of the gold standards in nursing education. In the world, eye tracking systems are used to determine the focal point. Eye tracking technology aims to record the movement of the eyeball to determine where the person is focusing while performing certain tasks. These systems have also contributed to the study of cognitive and neurological development. It has started to be used together with simulation training in health education. By determining where the student focuses during clinical practice simulation training using an eye tracker, it is possible to reschedule the practice training or to provide feedback on the student's misapplications during the application. The purpose of this research; The aim of this study is to develop an eye tracker for simulation training in nursing and to examine the effectiveness of an eye tracker in a simulation scenario.

DETAILED DESCRIPTION:
It is a double-blind randomized controlled experimental study in which two groups (experiment-control) will be compared and a post-test control group design will be used. The study consists of 2 stages. Stage 1: a) Developing the eye tracker, b) Preparing the simulation scenario and c) Conducting the pilot study. Stage 2: a) To examine the effectiveness of the developed eye tracker. To be included in the pilot study, it is necessary to be a 3rd year student of the nursing department, and to be a 4th year student of the nursing department to be included in the main application. 10 students will be included for the pilot study. The sample size was calculated in the G power statistics program by utilizing the data of a study in which on nursing students using a simulation intervention was previously performed (α =0.05, d=1.18). Accordingly, it was found that 13 people should be taken for each group to sampling for 80% power. Considering that there might be losses, the number of samples was increased by 10% and it was planned to include a total of 30 people in the study. Intention-to-treat analysis will be performed to manage bias and losses. After the eye tracker pilot application, eye tracker analysis data and video feedback data will be shared with students. Then, the personal information form to be used in the study, the simulation design scale, the student satisfaction and self-confidence scale in learning will be filled and analyzed. At the end of simulation, feedback will be received from the students participating in the pilot application Necessary changes will be made in the application simulation and eye tracker application in line with the feedback. Then the main application will be started. In the main application, eye tracker data and video feedback data will be shared with the experimental group students. Only video feedback data will be shared with the control group. In the main application, the forms and scales used in the pilot study will be used.

ELIGIBILITY:
Inclusion Criteria:

* To be a 3rd year student at Pamukkale University nursing department in order to be included in the pilot study.
* To be a 4th year student of Pamukkale University nursing department in order to be included in the main application.
* Not working as a nurse in any institution (high school/associate graduate nurse).
* Volunteer to participate in the study.

Exclusion Criteria:

* Not being a student of Pamukkale University nursing department (3rd year student for pilot study-4th year student for main application) on the specified dates.
* Working as a nurse in any institution (high school / associate degree nurse).
* Not volunteering to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Students' Satisfaction and Self-confidence Scale | up to 2 weeks
  This instrument is a 13-item scale used to measure student satisfaction with the simulation activity (5 items) and self-confidence in learning (8 items). Cronbach's alpha for satisfaction was 0.94; for self-confidence, it was 0.87. Responses are rated on a 5-point Likert scale with values ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher satisfaction and greater levels of selfconfidence.
Simulation Design Scale | up to 2 weeks
  The SDS is a 20-item tool developed to measure constructs from the Jeffries and Rizzolo (2006) simulation model. The design features rated by the students include objectives and information (five items), student support (four items), problem-solving (five items), guided reflection or feedback (four items), and fidelity (two items). Cronbach's alpha for the instrument was 0.92. Responses are rated on a 5-point Likert scale with values ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate increased recognition of design features in simulation.
Personal Information Form | up to 2 weeks
  The personal information form consists of a total of 9 questions about students' demographic information, reasons for choosing the nursing profession, and simulation experiences.

SECONDARY OUTCOMES:
Wound dressing checklist | up to 2 weeks
  It is a checklist developed by taking expert opinion on wound dressing. Before the study, students will be trained on wound dressing. This checklist will be used to assess students' proficiency in wound dressing application following the training provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydin Adnan Menderes Üniversitesi, Aydin, Turkey (Türkiye)